CLINICAL TRIAL: NCT05824481
Title: A Phase II Trial of Cadonilimab (AK104) Plus Lenvatinib in Patients With Advanced Endometrial Cancer
Brief Title: Study of Cadonilimab (AK104) Plus Lenvatinib in Patients With Advanced Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin Huang, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-099-01
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Endometrial Cancer; Endometrial Adenocarcinoma
Keywords: Endometrial Cancer; Immune Checkpoint Inhibitors (ICIs); Anti-PD-1/CTLA4 bi-specific antibody; Antiangiogenic agents; Lenvatinib
MeSH Terms: conditions — Endometrial Neoplasms | interventions — lenvatinib; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Intervention Model Description: Drug: Cadonilimab Drug: Lenvatinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab + Lenvatinib (Experimental): Safety run-in stage. A dose de-escalation schedule is used in this phase. Dose Level 1: cadonilimab 10 mg/kg administered intravenously on day 1 and lenvatinib 16 mg administered orally once daily on a 21-day treatment cycle. If ≥2/6 patients experience a DLT, we will de-escalate to Dose Level 2: cadonilimab 10 mg/kg administered intravenously on day 1 and lenvatinib 12 mg administered orally once daily on a 21-day treatment cycle. Approximately 3-12 patients will be enrolled in the safety run-in phase.
  Expansion stage. The expansion stage will begin once the RP2D of lenvatinib have been determined in the safety run-in phase in order to assess antitumor activity of cadonilimab and lenvatinib combination. In expansion stage, cadonilimab 10 mg/kg and lenvatinib PR2D will be administered.
  Interventions: Drug: Cadonilimab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Cadonilimab — Injectable solution
  Other Names: AK104
Drug: Lenvatinib — Capsule
  Other Names: Tyrosine Kinase Inhibitor

SUMMARY:
This is an open-label, multi-center Phase II study of cadonilimab (AK104) combined with lenvatinib in patients with advanced endometrial cancer. The primary objective is to evaluate objective response rate of cadonilimab plus lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF).
2. Has a histologically confirmed diagnosis of endometrial carcinoma (EC). Has documented evidence of metastatic or recurrent EC which is not amenable to curative treatment with surgery and/or radiation therapy.
3. Failure or intolerance of standard first-line platinum-based chemotherapy regimen for EC.

   Note: Prior adjuvant therapy is NOT counted as a systemic chemotherapeutic regimen for management of advanced EC. However, adjuvant chemotherapy could be counted as one prior regimen in patients who had recurrence during or within 12 months of completion of therapy. There is no restriction regarding hormonal therapy.
4. Age ≥ 18 years and ≤ 75 years.
5. Has measurable disease per RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Life expectancy exceeds 3 months.
8. Has adequate organ function as defined by the following criteria:

   * Absolute neutrophil count (ANC) (≥1.5×109/L), hemoglobin of ≥90 g/L, platelets ≥100 ×109/L
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN (however, patients with known liver metastasis who have AST or ALT level ≤ 5 × ULN may be enrolled)
   * Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula)

10. Women of childbearing potential should have a negative serum or urine pregnancy test prior to receiving the first dose of study treatment; and should be willing to use one acceptable contraception (i.e., oral contraceptives, condoms, intrauterine devices [IUDs]) throughout the period of taking study treatment and for at least 6 months after the last dose of study drug(s).

Exclusion Criteria:

1. Histologic types of carcinoma other than endometrial carcinoma.
2. Known or suspected allergy to any of study drugs.
3. Prior exposure to any anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, or small molecule anti-angiogenic agent.
4. Has an active autoimmune disease requiring systemic therapy (i.e., with use of disease modifying drugs, corticosteroids or immunosuppressive drugs) in past 2 years. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is permitted.
5. Concurrent medical condition requiring the use of systemic steroid therapy (dose >10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy within 2 weeks prior to the first dose of study intervention.
6. Has received anti-tumor treatment within 28 days, including but not limited to chemotherapy and radiotherapy or targeted therapy.
7. Any unresolved toxicities from prior therapy, greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment, with exception of alopecia and anemia.
8. Has an active infection requiring systemic therapy.
9. Clinically significant cardiovascular diseases, including but not limited to congestive heart failure (New York heart association [NYHA] class >2), unstable or severe angina, severe acute myocardial infarction within 6 months before enrollment, supraventricular or ventricular arrhythmia which need medical intervention, or QT interval male ≥ 450 ms, female ≥ 470 ms.
10. Hypertension that can not be well controlled through antihypertensive drugs (systolic pressure ≥140 mmHg and/or diastolic pressure ≥90 mmHg).
11. Received major surgery with 28 days before the first medication.
12. Coagulation abnormalities (INR >2.0, PT >16s), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
13. Proteinuria ≥ (++) or 24 hours total urine protein >1.0g.
14. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
15. Has known active hepatitis B disease (hepatitis B virus [HBV] DNA ≥1×104/ml) or hepatitis C disease (hepatitis C virus [HCV] RNA ≥1×103/ml).
16. History of another malignancy in the previous 3 years, with a disease-free interval of <3 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
17. Has known active central nervous system metastases.
18. Has a known history of immunodeficiency including human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease.
19. Has received a live vaccine within 30 days prior to the first dose of trial treatment. Note: Injection of inactivated viral vaccines against seasonal influenza are allowed.
20. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | the first 21 days of treatment
  MTD is defined as the highest dose level at which no more than 1 out of 6 subjects experiences a dose limiting toxicities (DLT) during the first cycle.
Recommended Phase 2 dose (RP2D) | the first 21 days of treatment
  Determine the RP2D of lenvatnib
Response Rate (ORR) | from the first drug administration up to two years
  ORR is the proportion of patients with best response of complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | from the first drug administration up to two years
  Proportion of patients whose best overall response is either CR, PR, or SD.
Duration of response (DOR) | from the first drug administration up to two years
  Time from first documented response (CR or PR) until documented disease progression or death, whichever occurs first.
Overall survival (OS) | from the first drug administration up to 2 years
  Time from the date of first study treatment administration to the date of death due to any cause.
Safety and tolerability | up to 90 days after last study treatment administration
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.

OTHER OUTCOMES:
Biomarkers associated with the response to cadonilimab plus lenvatinib | Samples taken prior to the first dose of drug, Cycle 3 and at progression
  Exploration of biomarkers that predict the efficacy of cadonilimab combined with lenvatinib

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Cetntre, Guangzhou, China